CLINICAL TRIAL: NCT04094116
Title: Comparison of Effectiveness of Ear Syringing With or Without Pre-Ear Oil Application , Non-randomized Control Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Chang Wells, resident, Hospital Authority, Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WON-20190902-11381
Record Dates: First submitted 2019-09-14; First posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Cerumen Impaction of Both Ears

STUDY DESIGN:
Intervention Model Description: non randomised control trials
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ear wax syringing with pre ear oil treatment (Active Comparator): patients in Fanling Family Medicine Centre with ear wax will be given ear oil one week before performing ear syringing.
  Interventions: Procedure: ear wax syringing without pre ear oil treatment
- ear wax syringing without pre ear oil treatment (Sham Comparator): Patients in Wong Siu Ching Clinic and Tai Po Clinic who are found to have ear wax after physical examination will have ear syringing done, without pre-ear oil application.
  Interventions: Procedure: ear wax syringing without pre ear oil treatment

INTERVENTIONS:
Procedure: ear wax syringing without pre ear oil treatment — Active Comparator: ear wax syringing with pre ear oil treatment Sham Comparator: ear wax syringing without pre ear oil treatment
  Other Names: ear wax syringing with pre ear oil treatment

SUMMARY:
Patients in Wong Siu Ching Clinic and Tai Po Clinic who are found to have ear wax after physical examination will have ear syringing done, without pre-ear oil application. On the other hand, patients in Fanling Family Medicine Centre with ear wax will be given ear oil one week before performing ear syringing. We will compare the respective success rates of ear syringing from these 2 groups, the mean numbers of syringing attempts , as well as any complications such as ear canal abrasion, ear drum perforation, any pain or vertigo reported by patients. For those cases who fail ear syringing , olive oil will be prescribe and arrange 1 week follow up for ear syringing .

DETAILED DESCRIPTION:
Patients in Wong Siu Ching Clinic and Tai Po Clinic who are found to have ear wax after physical examination will have ear syringing done, without pre-ear oil application. On the other hand, patients in Fanling Family Medicine Centre with ear wax will be given ear oil one week before performing ear syringing. We will compare the respective success rates of ear syringing from these 2 groups, the mean numbers of syringing attempts, subjective improvement in hearing , as well as any complications such as ear canal abrasion, ear drum perforation, any pain or vertigo reported by patients. For those cases who fail ear syringing , olive oil will be prescribe and arrange 1 week follow up for ear syringing .

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old, who complain about blocked ear found to have ear wax which impacts ear drum and able to sign consent.

Exclusion Criteria:

* Patients who are contraindicated to ear syringing will be excluded : otitis externa , otitis media , history of tympanic membrane perforation , history or ear surgery , unilateral deafness , in-co-operated patient (eg. Children ) , history of vertigo after ear syringing .

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The mean number of syringing attempts (50 ml syringe) | 1 day
  For both groups the mean number of syringing attempts (and 95% confidence interval) is calculated and compared by testing the difference between the means, using a t test for independent samples. For patients with persistent earwax in both ears , the mean number of syringing attempts needed for both ears in one patient is used for the calculations . All ears in which the wax is still persistent after another 10 syringing attempts are given a value of 11 in the calculations . Data for this study is analyzed using SPSS version 26 .

SECONDARY OUTCOMES:
The presence of ear canal abrasion, | 1 month
  The presence of ear canal abrasion,

CONTACTS AND LOCATIONS:
Locations (3):
- Hong Kong (3):
  - Fanling Family MEdicine Centre , 1/F , 2 , Pik Fung Road , Fan Ling, Hong Kong
  - Tai Po Jockey Club Clinic , 37 Ting Kok Road , Tai Po , Hong Kong, Hong Kong
  - Wong Siu Ching Family Medicine centre . 1 , Po Wu Lane , Tai Po, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eekhof JA, de Bock GH, Le Cessie S, Springer MP. A quasi-randomised controlled trial of water as a quick softening agent of persistent earwax in general practice. Br J Gen Pract. 2001 Aug;51(469):635-7. PMID 11510392
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/11510392